CLINICAL TRIAL: NCT00357591
Title: MOMENTUM: Multicenter Trial of the Orqis Medical CRS for the Enhanced Treatment of CHF Unresponsive to Medical Therapy
Brief Title: Randomized Trial for Patients With Chronic Heart Failure With Acute Decompensation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Projected neutral significance for primary composite efficacy endpoint.
Sponsor: Orqis Medical Corporation (Industry)
Responsible Party: Irene Parker/VP Regulatory Affairs, Orqis Medical Corporation
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IDEG020301
Record Dates: First submitted 2006-07-25; First posted 2006-07-27 (Estimated); Last update posted 2009-12-25 (Estimated); Status verified 2009-08

CONDITIONS: Heart Failure, Congestive
Keywords: Heart Failure; Acute Decompensation; Chronic Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Control (Active Comparator)
  Interventions: Device: Continuous Aortic Flow Augmentation

INTERVENTIONS:
Device: Continuous Aortic Flow Augmentation — 1.0-1.5 lpm augmented blood flow

SUMMARY:
The Company's proprietary products are based on Orqis Medical's hypothesis, supported by early clinical data, that increasing and maintaining continuous blood flow in the descending aorta, known as continuous aortic flow augmentation or CAFA, improves hemodynamics in heart failure patients. The clinical impact of the hemodynamic improvement is currently being evaluated to determine the effects of CAFA on stopping or reversing the progression of heart failure through three physiological effects:

* VASCULAR - Reducing systemic vascular resistance
* RENAL - Improving renal function
* CARDIAC - Reducing cardiac workload

ELIGIBILITY:
Inclusion Criteria:

1. Patients hospitalized due to decompensated heart failure who require IV inotropic and/or vasodilator and diuretic therapy
2. Patients receiving appropriate medical therapy for heart failure, defined as ACE inhibitors and beta blockers (all unless not tolerated or contraindicated) and diuretics, for 1 month prior to study entry
3. For at least 24 hours prior to inclusion into the study, the patient should be treated with a minimum dose of the following: dobutamine 2.5μg/kg/min or milrinone 0.3μg/kg/min or dopamine 5μg/kg/min. or nesiritide 0.01μg/kg/min or nitroglycerin 0.3 µg/kg/min or nitroprusside 0.3 µg/kg/min or a combination of any of these agents, with diuretic therapy. Doses of the above stated medications should be stable for 6 hours prior to inclusion into study. An increase in this dosage within the first 8 hours after enrollment is determined by the attending physician to be unlikely and the following definition of "not responding adequately to IV inotropic and/or vasodilator and diuretic therapy" is exhibited:

   * PCWP is ≥ 20 mmHg at time of randomization and PCWP was ≥ 18 mmHg continuously for 24 hours or PCWP ≥ 20 mmHg continuously for 12 hours prior to randomization.
   * Cardiac Index < 2.4 L/min/m2
   * There is evidence for abnormal renal function and/or diuretic resistance defined as: Serum creatinine > 1.2 mg/dL or Diuretic dosage of intravenous Furosemide ≥ 120 mg daily, or equivalent
4. LVEF < 35%
5. Male or female 18-90 years of age
6. If female, no child-bearing potential or negative pregnancy test
7. Written informed consent
8. Willingness to participate in required follow-up exams

Exclusion Criteria:

1. Acute Q-wave myocardial infarction within past 7 days
2. Post cardiotomy shock within past 30 days
3. Cardiac surgery within past 14 days
4. Bridge to transplant
5. History of severe COPD as defined as FEV1 < 1.0 liter
6. History of malignant arrhythmias defined as either:

   * sustained ventricular tachycardia > 15 beats or more in length, not associated with a correctable cause, within the preceding 3 months, unless the patient presently has an implantable cardiac defibrillator.
   * history of ventricular fibrillation or sudden death, unless the patient presently has an implantable cardiac defibrillator
7. Patients implanted with a resynchronization device within the previous 14 days or if there is a possibility of implant within 60 days following randomization
8. Systolic pressure <80 mmHg
9. Requiring cardiopulmonary support type devices
10. Platelets < 50,000/mm3 or other evidence of coagulopathy, INR greater than 1.5 in the absence of anticoagulation therapy.
11. Infection (WBC ≥ 12.5 x 103/ml, and or temperature ≥ 100.5°F/38°C)
12. History of cerebral vascular accident (CVA) or transient ischemic attacks (TIA) within the last 3 months
13. Unwilling or unable to receive blood transfusion
14. Inability to undergo treatment with heparin
15. Patients on dialysis or serum creatinine > 4.0 mg/dl
16. Primary liver disease with bilirubin, SGOT, or SGPT > 4X upper limit of normal
17. Life expectancy from other disease < 12 months
18. Patients who are active on the cardiac transplantation waiting list, unless there is a documented reason (large body habitus, highly sensitized, O blood group) to anticipate that transplant is unlikely within the subsequent 65 days.
19. Symptomatic patent foramen ovale or intracardiac shunt
20. Patients diagnosed with clinically significant peripheral vascular disease, defined as absent pedal pulse or signs or symptoms of limb ischemia, including a history of intermittent claudication
21. Patients with amyloidosis, thyroid induced heart failure, high output failure secondary to an arterio-venous fistula, and significant uncorrected primary valvular disease (with the exception of mitral regurgitation believed secondary to LV dilatation)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2004-09; Primary Completion 2008-01 (Estimated); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Alive, Number of days out of the hospital, not on mechanical assistance over 35 day period. | 35 days

CONTACTS AND LOCATIONS:
Overall Officials: Barry H Greenberg, M.D., Principal Investigator — University of California, San Diego
Locations (1):
- University of California at San Diego, San Diego, California, United States

REFERENCES:
- [Derived] Zile MR, Colombo PC, Mehra M, Greenberg B, Brown S, Konstam MA. Progressive improvement in cardiac performance with continuous aortic flow augmentation (aortic flow therapy) in patients hospitalized with severe heart failure: results of the Multicenter Trial of the Orqis Medical Cancion System for the Enhanced Treatment of Heart Failure Unresponsive to Medical Therapy (MOMENTUM). J Heart Lung Transplant. 2010 Jan;29(1):86-92. doi: 10.1016/j.healun.2009.10.005. PMID 20123246
- [Derived] Greenberg B, Czerska B, Delgado RM, Bourge R, Zile MR, Silver M, Klapholz M, Haeusslein E, Mehra MR, Mather P, Abraham WT, Neaton JD, Brown BS, Parker IC, Konstam MA; MOMENTUM Investigators and Coordinators. Effects of continuous aortic flow augmentation in patients with exacerbation of heart failure inadequately responsive to medical therapy: results of the Multicenter Trial of the Orqis Medical Cancion System for the Enhanced Treatment of Heart Failure Unresponsive to Medical Therapy (MOMENTUM). Circulation. 2008 Sep 16;118(12):1241-9. doi: 10.1161/CIRCULATIONAHA.108.773275. Epub 2008 Sep 2. PMID 18765394